CLINICAL TRIAL: NCT01673529
Title: A Two Part Randomized, Double-blind, Placebo Controlled Study to Investigate the Effects of Topical Doses of SB705498 Oncapsaicin, Histamine, and Cowhage Responses in Healthy Volunteers.
Brief Title: Investigation of Topical SB705498 on Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115246
Record Dates: First submitted 2012-07-12; First posted 2012-08-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Dermatitis, Atopic
Keywords: Pruritus; TRPV1; Cowhage; Atopic Dermatitis; Capsaicin; Itch; Histamine; healthy volunteers; SB705498; Clinical
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- study population (Experimental): All subjects will receive 1%, 3%, 5% (w/w) of SB705498 and a placebo comparator
  Interventions: Drug: SB705498; Drug: Placebo

INTERVENTIONS:
Drug: SB705498 — 1%, 3% and 5% (w/w) of SB705498 will be used in part A of the study. One dose will then be selected based on criteria explained in the protocol for use in Part B of the study.
Drug: Placebo — Placebo to match SB705498 will be used in both Part A and Part B of the study.

SUMMARY:
A two part, randomized, double-blind, placebo controlled study to investigate the effects of topical doses of SB705498 in healthy volunteers.

DETAILED DESCRIPTION:
This study is a two part, randomized, double-blind, placebo controlled study to investigate the effects of topical doses of SB705498 on capsaicin, histamine, and cowhage responses in healthy volunteers. Part A has been designed to establish whether the topical formulation is capable of delivering SB705498 to the proposed site of action, and to select an appropriate dose for Part B. Part B will examine the effects of SB705498 on pruritus initiated by a histaminergic and a non-histaminergic pathway, using two different challenge agents; histamine and cowhage. This may provide important information about the role of TRPV1 in pruritus and the therapeutic potential of SB705498.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian volunteers aged between 18 and 65 years of age inclusive, at time of signing the informed consent. Healthy subjects are defined as individuals who are not taking any regular medication and are free from clinically significant illness or disease as determined by their medical history (including family history), physical examination, 12-lead ECG, laboratory studies, and other tests specified in this protocol.
* Subject has the ability to read, comprehend, and record information required by protocol, and is willing and able to provide signed and dated written informed consent prior to study participation, including compliance with the requirements and restrictions listed in the consent form.
* Non smoker who has not smoked or used nicotine containing products for a minimum period of 6 months prior to the screening visit.
* Subject must score greater than 40 on a COVAS scale of 0-100 for itch induced by both cowhage and histamine at screening and show a flare response with capsaicin measured by LDI scan.
* Is willing to avoid UV exposure. i.e. use of Sun beds and sunbathing for 7 days prior to screening, throughout the study and and until a week after the last dose. Subjects who require treatment with photosensitizing drugs (e.g, tetracycline, thiazides, fluoroquinolones, phenothiazines, or sulfonamides) will withdrawn. Subjects must also be willing to use sunscreen of SPF30 or above on the volar surface of the forearms for a week after the last dose.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 MlU/ml and estradiol less than 40 pg/ml (less than 147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in the protocol if they wish to continue their HRT during the study.

Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.]; Child-bearing potential and agrees to use one of the contraception methods listed in the protocol. Female subjects willing to participate in the study must agree to use contraception from the screening visit until 15 days post-last treatment administration.

* Male subjects must agree to use one of the contraception methods listed in the protocol. For male subjects willing to participate in the study this criterion must be followed from the time of the screening visit until 15 days post-last treatment
* BMI within the range 19.0 - 32.0 kg/m2 (inclusive).
* AST and ALT less than 2xULN; alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin.
* QTcB or QTcF less than 450 msec. Note that if the initial QTc value is prolonged, the ECG should be repeated two more times (with 5 minutes between ECG readings) and the average of the three QTc values used to determine eligibility.

Exclusion Criteria:

* Suffers from skin infection or inflammation of the forearm, or has other arm skin irregularities that may in the opinion of the investigator interfere with study assessments (e.g. nevi, tattoos).
* The subject suffers from eczema, psoriasis or any other acute or chronic dermatological problem if, in the opinion of the investigator this is likely to interfere with study assessments
* Any subject with localised sunburn in the area to be treated as part of the study.
* History of regular alcohol/drug consumption within 6 months of the study. Regular alcohol consumption defined as: an average weekly intake of greater than 21 units for males and greater than 14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, one glass (125 ml) of wine or one (25 ml) measure of spirits.
* A positive pre-study drug/alcohol screen at screening visit. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial resulting in exposure to more than four new chemical entities within 12 months prior to the first dosing day or has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unable to refrain from use of prescription or non-prescription drugs. Refer to the protocol for details.
* History of sensitivity to any of the study medications SB705498, challenge agents or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period following completion of the study.
* Lactating females.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for HIV antibody.
* Excessive caffeine drinkers (approximately 5 or more cups a day) or the subject is unable to commit to refraining from caffeine-containing products for 24hrs prior to each assessment visit and whilst present in the unit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07-17 (Actual); Primary Completion 2012-10-04 (Actual); Study Completion 2012-10-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the area of flare induced by capsaicin as assessed by Laser | 1 hour
2) Average itch over maximum of 15 minutes post application of challenge agent | 15 minutes

SECONDARY OUTCOMES:
vital sign measurements, ECG, Clinical Laboratory data and Adverse Events | 3 months
  safety and tolerability
Peak itch intensity on 0 to 100 COVAS (Computerised visual analogue scale) | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Gibson RA, Robertson J, Mistry H, McCallum S, Fernando D, Wyres M, Yosipovitch G. A randomised trial evaluating the effects of the TRPV1 antagonist SB705498 on pruritus induced by histamine, and cowhage challenge in healthy volunteers. PLoS One. 2014 Jul 21;9(7):e100610. doi: 10.1371/journal.pone.0100610. eCollection 2014. PMID 25047038
- See also: Results for study 115246 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115246?search=study&study_ids=115246#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115246 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register